CLINICAL TRIAL: NCT01656317
Title: Effect of Early Rehabilitation in Patients With Acute Subarachnoid Hemorrhage
Brief Title: Rehabilitation of Patients After Subarachnoid Hemorrhage
Acronym: SAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Tanja Karic, medical doctor, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/2189.; ID:2011/2189. (Other Grant/Funding Number: Oslo University Hospital)
Record Dates: First submitted 2012-07-12; First posted 2012-08-02 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: SAH
Keywords: SAH; Early rehabilitation; Mobilisation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilisation of patients after SAH (Active Comparator): Patients which were treated after SAH in 2012 will receive early multidisciplinary rehabilitation consist of individualized stimulation and mobilisation.
  Mobilisation will be initiated and completed according to mobilisations guidelines which are developed and adjusted to the patients in early stage after aneurysmal SAH.
  Interventions: Other: Early multidisciplinary rehabilitation
- Patients after SAH from 2011 (No Intervention): Patients after SAH from 2011 which did not receive early rehabilitation and mobilisation will be followed up 3-6 annd 12 months after SAH and outcome measures compared with patients from 2011.

INTERVENTIONS:
Other: Early multidisciplinary rehabilitation — Multidisciplinary rehabilitation consist of individualized stimulation and mobilisation.
  The multidisciplinary team consists of a physician, a nurse, a physiotherapist, an occupational therapist and a clinical neuropsychologist.
  Arms: Mobilisation of patients after SAH

SUMMARY:
The study's main objective will be to assess which effect early initiated rehabilitation has on the frequency of complications and the level of physical and cognitive functioning after aneurysmal subarachnoid hemorrhage (SAH).

To this end the following aspects will be investigated:

The frequency of complications (with special emphasis on pulmonary complications,thromboembolic events, cerebral vasospasm, unintended discontinuation of drains and lines)

* Length of stay in hospitals and socio-economic impact
* Physical and cognitive function in the early and chronic phase after SAH
* Health-related quality of life and participation in society in the chronic phase

DETAILED DESCRIPTION:
Oslo University Hospital (OUS) is the primary hospital for Health Region South-East regarding treatment of patients with SAH. Approximately 120 patients are referred annually. OUS,Rikshospitalet, Dept of Neurosurgery offers 24/7 service of surgical and vascular aneurysm repair performed by a dedicated vascular team.

Patients admitted in 2012 are treated in accordance to the standard institutional protocol plus an early rehabilitation model adapted to SAH, while patients admitted in 2011 who did not receive any early rehabilitation, but apart from that were treated identically, serve as a control group.

All patients admitted to the intermediate unit at OUS in 2011 and 2012 with aneurysmal SAH and repaired aneurysm will be invited to participate in this study. Examination of the patients from both 2011 and 2012 will be performed as part of routine, neurosurgical follow- up which is in the early phase at 3-6 months and in the chronic phase at least 12 months post SAH. Exclusion criteria for participation in the study: unsecured ruptured aneurysm, symptomatic aneurysm without rupture, previous SAH or brain injury, diagnosis of a neurodegenerative disorder, patients from other health regions or tourists, patients that were treated at the intensive care unit (ICU )only.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the intermediate unit at OUS in 2011 and 2012 with aneurysmal SAH and repaired aneurysm will be invited to participate in this study.

Exclusion Criteria:

* Unsecured ruptured aneurysm,
* Symptomatic aneurysm without rupture
* Previous SAH or brain injury, diagnosis of a neurodegenerative disorder
* Patients from other health regions or tourists
* Patients that were treated at the intensive care unit (ICU )only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-02-27 (Actual); Study Completion 2015-12-20 (Actual)

PRIMARY OUTCOMES:
Glasgow Coma Scale (GCS) | up to 10 weeks

SECONDARY OUTCOMES:
Glasgow Outcome Scale Extended (GOSE) | 3-6 months and 12 months after SAH
Functional Independence Measure (FIM) | 3-6 months and 12 months after SAH
Coma Recovery Scale (CRS) | 3-6 and 12 months after SAH
Disability Rating Scale (DRS) | 3-6 and 12 months after SAH
High Level Mobility Assessment Tool (HIMAT) | 3-6 and 12 months after SAH

OTHER OUTCOMES:
Pain score on the Visual Analog Scale | 3-6 and 12 months after SAH

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Karic, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Karic T, Roe C, Nordenmark TH, Becker F, Sorteberg W, Sorteberg A. Effect of early mobilization and rehabilitation on complications in aneurysmal subarachnoid hemorrhage. J Neurosurg. 2017 Feb;126(2):518-526. doi: 10.3171/2015.12.JNS151744. Epub 2016 Apr 8. PMID 27058204
- Available data/document: Article: DOI: 10.2340/16501977-2121 — https://www.ncbi.nlm.nih.gov/pubmed/27494170 — Impact of early mobilization and rehabilitation on global functional outcome one year after aneurysmal subarachnoid hemorrhage. Karic T1,2, Røe C1,3, Nordenmark TH1, Becker F4,3, Sorteberg W2, Sorteberg A2,3.
- Available data/document: Article: DOI: 10.3171/2015.12.JNS151744 — https://www.ncbi.nlm.nih.gov/pubmed/27058204 — J Neurosurg. 2017 Feb;126(2):518-526. doi: 10.3171/2015.12.JNS151744. Epub 2016 Apr 8. Effect of early mobilization and rehabilitation on complications in aneurysmal subarachnoid hemorrhage. Karic T1,2, Røe C1,3, Nordenmark TH1, Becker F4,3, Sorteberg W2, Sorteberg A2,3.
- Available data/document: Article: 10.3109/09638288.2014.966162 — https://www.ncbi.nlm.nih.gov/pubmed/25264735 — Disabil Rehabil. 2015;37(16):1446-54. doi: 10.3109/09638288.2014.966162. Epub 2014 Sep 29. Early rehabilitation in patients with acute aneurysmal subarachnoid hemorrhage. Karic T1, Sorteberg A, Haug Nordenmark T, Becker F, Roe C.